CLINICAL TRIAL: NCT01723475
Title: An Open-label, Phase I, Dose-escalation Study to Characterize the Safety, Tolerability, Pharmacokinetics, and Maximum Tolerated Dose of BAY 2010112, Given Once Daily by Subcutaneous Administration or by Continuous Intravenous Infusion, in Subjects With Castration-resistant Prostate Cancer
Brief Title: First-in-man Dose Escalation Study of BAY2010112 in Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15590; 2012-000691-42 (EudraCT Number)
Record Dates: First submitted 2012-11-01; First posted 2012-11-08 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Prostatic Neoplasms
Keywords: Phase I; Dose Escalation; Prostate cancer; Antibodies; Bispecific T-cell Engager (BiTE)
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAY2010112 (s.c.) (Experimental)
  Interventions: Biological: BAY2010112
- BAY2010112 (c.i.v.) (Experimental)
  Interventions: Biological: BAY2010112

INTERVENTIONS:
Biological: BAY2010112 — Subcutaneous (s.c.) administration once daily. Starting dose will be 0.5 µg ; dose will be escalated dependent on any dose limiting toxicities
  Arms: BAY2010112 (s.c.)
Biological: BAY2010112 — Continuous intravenous infusion (c.i.v.) administration. Starting dose will be 5 µg ; dose will be escalated dependent on any dose limiting toxicities.
  Arms: BAY2010112 (c.i.v.)

SUMMARY:
This is the first study where BAY2010112 is given to humans. Patients with castration resistant prostate cancer will be treated. Every patient will receive drug treatment, there is no placebo group. Patients will receive different dosages of BAY2010112 to determine the safety, tolerability and maximum tolerated dose (MTD) of BAY2010112.

The study will also assess the pharmacokinetics and the clinical efficacy of BAY2010112.

BAY2010112 will be given daily as subcutaneous injection or as continuous intravenous infusion. Treatment will be stopped if the tumor continues to grow, if side effects, which the patient cannot tolerate, occur or if the patient decides to exit treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects, aged >/= 18 years
* Subjects with histologically or cytologically proven advanced castration-resistant prostate cancer (CRPC)

  * who failed at least 1 taxane regimen and are refractory to abiraterone and/or enzalutamide therapy OR
  * who have actively refused any treatment which would be regarded standard.
* Subjects should have undergone bilateral orchiectomy or should be on continuous androgen deprivation therapy with a gonadotropin releasing hormone agonist or antagonist.
* Subjects must have shown progressive disease after discontinuation of anti-androgen therapy (i.e. flutamide, bicalutamide or nilutamide) before study drug treatment.
* Total serum testosterone should be less than 50 ng/ml or 1.7 nmol/L
* Evidence of progressive disease, defined as one or more (Prostate Cancer Working Group 2 (PCWG2) criteria):
* PSA level of at least 2 ng/ml that has risen on at least 2 successive occasions at least 1 week apart
* Nodal (in lymph nodes >/= 2cm) or visceral progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST)
* Appearance of one more new lesions in bone scan
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
* Life expectancy of at least 3 months

Exclusion Criteria:

* Any anticancer therapy or immunotherapy within 4 weeks of start of first dose
* Confirmed history or current autoimmune disease or other diseases resulting in permanent immunosuppression or requiring permanent immunosuppressive therapy
* Prior radiotherapy (local palliative radiotherapy is permitted)
* History of allergic reactions to monoclonal antibody therapy
* History of clinical significant cardiac disease: including unstable angina, acute myocardial infarction within 6 months prior to first study treatment, congestive heart failure ≥New York Heart Association (NYHA) Class III), and arrhythmia requiring therapy except for beta-blockers, calcium channel blockers and digoxin or uncontrolled hypertension, despite optimal medical management
* Clinically relevant findings in the electrocardiogram (ECG) such as a second- or third-degree AV block, prolongation of the QRS complex over 120 msec or of the QT interval corrected for heart rate (QTc)-interval over 450 msec
* Current evidence or history of uncured (i.a. any absolute risk of latent infection) of hepatitis B or C or human immunodeficiency virus (HIV) infection
* Chronic systemic corticosteroid therapy or any other immunosuppressive therapies should have been stopped at screening start
* Seizure disorder requiring therapy (such as steroids or anti-epileptics)
* Subjects unable to inject the study drug subcutaneously for intended s.c. application
* Non-suitable for a central venous access for intended c.i.v. administration

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-11-02 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events as a Measure of Safety and Tolerability | Up to 2 years or longer if indicated
Maximum Tolerated Dose (MTD) | Up to 2 years or longer if indicated
  MTD is measured by adverse event profile at the end of Cycle 1. MTD will be the highest dose level achieved during dose escalation where the incidence of dose-limiting toxicities (DLTs) is below 20%

SECONDARY OUTCOMES:
Maximum drug concentration (Cmax) of BAY2010112 in serum after single and multiple doses administration | Cycle 1 Day1 and 15; (1 Cycle is 21 days long)
Area under the concentration versus time curve (AUC) from zero to infinity after single (first) and multiple doses of BAY2010112 | Cycle 1 (1 Cycle is 21 days long)
Tumor response | Up to 2 years or longer if indicated
  Tumor response is measured by measurable lesions
Prostate-specific antigen (PSA) response | Up to 2 years or longer if indicated
  PSA response is measured by maximum decline in PSA that occurs at any point after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (5):
- Austria (2):
  - Linz, Upper Austria
  - Vienna
- Germany (3):
  - Heidelberg, Baden-Wurttemberg
  - Würzburg, Bavaria
  - Berlin

REFERENCES:
- [Result] Frankel SR, Baeuerle PA. Targeting T cells to tumor cells using bispecific antibodies. Curr Opin Chem Biol. 2013 Jun;17(3):385-92. doi: 10.1016/j.cbpa.2013.03.029. Epub 2013 Apr 25. PMID 23623807
- [Derived] Penny HL, Hainline K, Theoharis N, Wu B, Brandl C, Webhofer C, McComb M, Wittemer-Rump S, Koca G, Stienen S, Bargou RC, Hummel HD, Loidl W, Grullich C, Eggert T, Tran B, Mytych DT. Characterization and root cause analysis of immunogenicity to pasotuxizumab (AMG 212), a prostate-specific membrane antigen-targeting bispecific T-cell engager therapy. Front Immunol. 2023 Oct 23;14:1261070. doi: 10.3389/fimmu.2023.1261070. eCollection 2023. PMID 37942314
- [Derived] Hummel HD, Kufer P, Grullich C, Seggewiss-Bernhardt R, Deschler-Baier B, Chatterjee M, Goebeler ME, Miller K, de Santis M, Loidl W, Dittrich C, Buck A, Lapa C, Thurner A, Wittemer-Rump S, Koca G, Boix O, Docke WD, Finnern R, Kusi H, Ajavon-Hartmann A, Stienen S, Sayehli CM, Polat B, Bargou RC. Pasotuxizumab, a BiTE(R) immune therapy for castration-resistant prostate cancer: Phase I, dose-escalation study findings. Immunotherapy. 2021 Feb;13(2):125-141. doi: 10.2217/imt-2020-0256. Epub 2020 Nov 10. PMID 33172323
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/